CLINICAL TRIAL: NCT04657198
Title: A Phase 2b, Open-label, Multi-center, Extension Study to Evaluate the Safety and Immunogenicity of a Revaccination Dose of the RSVPreF3 Older Adults (OA) Investigational Vaccine Administered Intramuscularly 18 Months Post-Dose 2 in Adults 60 Years and Older Who Participated in the RSV OA=ADJ-002 Study
Brief Title: Extension Study to Evaluate the Safety and Immunogenicity of a Revaccination Dose of the RSVPreF3 OA Investigational Vaccine in Adults 60 Years and Older Who Participated in the RSV OA=ADJ-002 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 213569; 2020-000692-21 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: This is an open-label study, as all participants will receive the same RSVPreF3 OA investigational vaccine. No blind is used. Both the investigator and the participant know the identity of the intervention assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group High Dose_Adjuvanted (Experimental): Participants in one of the high dose adjuvanted groups in part B of the parent study RSV OA=ADJ-002: Group High Dose Adjuvanted will receive one revaccination dose of the RSVPreF3 OA investigational vaccine in the current study by intramuscular (IM) injection in the non-dominant arm.
  Interventions: Biological: RSVPreF3 OA investigational vaccine (GSK3844766A)
- Group Medium Dose_Adjuvanted (Experimental): Participants in one of the medium dose adjuvanted groups in part B of the parent study RSV OA=ADJ-002: Group Medium Dose Adjuvanted will receive one revaccination dose of the RSVPreF3 OA investigational vaccine in the current study by IM injection in the non-dominant arm.
  Interventions: Biological: RSVPreF3 OA investigational vaccine (GSK3844766A)
- Group Low Dose_Adjuvanted (Experimental): Participants in one of the low dose adjuvanted groups in part B of the parent study RSV OA=ADJ-002: Group Low Dose Adjuvanted will receive one revaccination dose of the RSVPreF3 OA investigational vaccine in the current study by IM injection in the non-dominant arm.
  Interventions: Biological: RSVPreF3 OA investigational vaccine (GSK3844766A)

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine (GSK3844766A) — RSVPreF3 OA investigational vaccine administered intramuscularly in the deltoid region of the non-dominant arm, at Day 1 (18 months post-Dose 2 in the RSV OA=ADJ-002 parent study).

SUMMARY:
Nine different formulations of the RSVPreF3 OA investigational vaccine were tested in the parent study (NCT03814590). Based on safety and immunogenicity data from the parent study, RSVPreF3 OA investigational vaccine will be evaluated in further clinical research. Participants in selected groups will be invited to participate in this extension study. All participants who will be enrolled in the current extension study will receive the RSV investigational vaccine approximately 18 months after they received their respective dose-2 in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, who received 2 doses of RSVPreF3 OA investigational vaccine and formulations with matched adjuvant in part B of the parent study RSV OA=ADJ-002: recombinant RSVPreF3 antigen doses of low, medium and high strengths with adjuvant.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for the follow-up visit, be available for contact)
* Written informed consent obtained from the participant prior to performance of any study specific procedure.

Exclusion Criteria:

Medical conditions

* Significant underlying illness or administered therapy that in the opinion of the investigator would be expected to prevent participation in the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on information on concomitant medication/vaccination collected prior to the study start and physical examination.
* Serious or unstable chronic illness that developed during or after the parent study. Patients with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as clinically stable.
* Recurrent or un-controlled neurological disorders or seizures that developed during or after the parent study. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that developed during or after the parent study, that in the opinion of the investigator would be expected to prevent completion of the study.
* Lymphoproliferative disorder and malignancy developed during or after the parent study.
* Any medical condition that developed during or after the parent study, that in the judgment of the investigator would make intramuscular injection unsafe.
* Previous vaccination with RSV vaccine, other than the one in the parent study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccine during the period beginning 30 days before the dose of study vaccine, or planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after the dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after the study vaccination.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the vaccine dose or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Confirmed use or anticipated use of immunosuppressive/cytotoxic therapy.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other exclusions

* Bedridden participants.
* Planned move to a location that will prohibit participating in the trial.
* History of chronic alcohol consumption and/or drug abuse that developed during or after the parent study as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, San Antonio, Texas
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Leroux-Roels I, Van Ranst M, Vandermeulen C, Abeele CV, De Schrevel N, Salaun B, Verheust C, David MP, Kotb S, Hulstrom V. Safety and Immunogenicity of a Revaccination With a Respiratory Syncytial Virus Prefusion F Vaccine in Older Adults: A Phase 2b Study. J Infect Dis. 2024 Feb 14;229(2):355-366. doi: 10.1093/infdis/jiad321. PMID 37699064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From a total of 126 participants enrolled in this study, 4 participants were withdrawn before vaccination. 122 participants received the study vaccination.
Groups:
- High Dose_AS01E Group: Participants received 1 dose of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E in the current study after having received 2 doses of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E in the RSV OA=ADJ-002 (NCT03814590) parent study.
- Low Dose_AS01E Group: Participants received 1 dose of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E in the current study after having received 2 doses of the RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01E in the RSV OA=ADJ-002 (NCT03814590) parent study.
- Medium Dose_AS01E Group: Participants received 1 dose of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E in the current study after having received 2 doses of the RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01E in the RSV OA=ADJ-002 (NCT03814590) parent study.
Period: Overall Study
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Started | 40 | 39 | 43
Completed | 39 | 39 | 43
Not Completed | 1 | 0 | 0
Not completed — CONSENT WITHDRAWAL, NOT DUE TO A (S)AE | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group | Total
Number analyzed (Participants) | 40 | 39 | 43 | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (5.4) | 69.1 (5.3) | 66.6 (5.6) | 68.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 24 | 72
  Male | 13 | 18 | 19 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 1 | 0 | 0 | 1
  Black Or African American | 1 | 2 | 1 | 4
  White | 38 | 37 | 42 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Solicited Administration Site Adverse Events (AEs)
Description: Assessed solicited administration site AEs are erythema, pain and swelling. Any pain is defined as any pain regardless of intensity grade. Any injection site erythema/swelling is scored with a diameter larger than (>) 20 millimeters (mm).
Time Frame: During the 4-day follow-up period post-vaccination (i.e. on the day of vaccination [Day 1] and 3 subsequent days)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants
  Any erythema | 1 | 6 | 5
  Any pain | 21 | 23 | 26
  Any swelling | 0 | 2 | 4

2. Primary Outcome: Number of Participants With Any Solicited Systemic AEs
Description: Assessed solicited systemic AE is fever (any temperature greater than or equal to 38.0 °C - the preferred location for measuring temperature being the oral cavity). Any is defined as occurrence of the symptom regardless of intensity grade or relation to study.
Time Frame: During the 4-day follow-up period post-vaccination (i.e. on the day of vaccination [Day 1] and 3 subsequent days)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 1 | 1 | 4

3. Primary Outcome: Number of Participants With Any Unsolicited AEs
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited AE. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 30-day follow-up period post-vaccination (i.e., on the day of vaccination [Day 1] and 29 subsequent days)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 5 | 11 | 12

4. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) up to 30 Days Post-vaccination
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity. Any is defined as any occurrence of SAE regardless of intensity grade or relation to study vaccination.
Time Frame: From Day 1 up to 30 days post-vaccination (Day 31)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Any Potential Immune-mediated Diseases (pIMDs) up to 30 Days Post-vaccination
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any is defined as the occurrence of any pIMD regardless of intensity grade or relation to study vaccination.
Time Frame: From Day 1 up to 30 days post-vaccination (Day 31)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 0 | 0 | 0

6. Primary Outcome: Humoral Immune Response in Terms of Neutralizing Antibody Titers Against Respiratory Syncytial Virus (RSV)-Serotype A
Description: Serological assays for the determination of functional antibodies against RSV-A are performed by neutralization assay. Anti RSV-A neutralizing antibody titers are given as Geometric Mean Titers (GMTs) and expressed as Estimated Dose: serum dilution giving a 60% reduction of the signal compared to a control without serum (ED60).
Time Frame: At 30 days post-vaccination (Day 31)
Population: The analysis was performed on the Per Protocol Set (that included participants who received the study intervention dose and have post-vaccination data, minus participants with protocol deviations that led to exclusion), for the High Dose_AS01E Group only (as per protocol).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | High Dose_AS01E Group
Number analyzed (Participants) | 34
Titers | 4394.9 [3191.3 to 6052.5]

7. Primary Outcome: Humoral Immune Response in Terms of Neutralizing Antibody Titers Against RSV-serotype B
Description: Serological assays for the determination of functional antibodies against RSV-B are performed by neutralization assay. Anti RSV-B neutralizing antibody titers are given as GMTs and expressed as ED60.
Time Frame: At 30 days post-vaccination (Day 31)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | High Dose_AS01E Group
Number analyzed (Participants) | 34
Titers | 6094.3 [4476.8 to 8296.4]

8. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3-specific Immunoglobulin G (IgG) Antibody Concentrations
Description: The detection and the quantification of total IgG antibodies directed against RSVPreF3 in human serum samples were based on an indirect Enzyme-Linked Immunosorbent Assay (ELISA). Anti RSVPreF3 antibody concentration is given in geometric mean concentration (GMC) and is expressed in ELISA Laboratory Units per milliliter (ELU/mL).
Time Frame: At 30 days post-vaccination (Day 31)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | High Dose_AS01E Group
Number analyzed (Participants) | 34
ELU/mL | 46276.5 [36821.3 to 58159.6]

9. Secondary Outcome: Frequency of RSVPreF3-specific Cluster of Differentiation 4+ (CD4+) T-cells Identified as Expressing at Least Two Markers
Description: Among markers expressed are interleukin-2 (IL2), cluster of 40 ligand (CD40L), tumour necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At 30 days post-vaccination (Day 31)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cells per million CD4+ T Cells
Arm/Group | High Dose_AS01E Group
Number analyzed (Participants) | 31
cells per million CD4+ T Cells | 1601 [1174 to 2541]

10. Secondary Outcome: Number of Participants With Any SAEs, up the End of Follow-up Study Period (Month 6)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity.
Time Frame: From Day 1 up to the end of follow-up period (Month 6)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 1 | 1 | 2

11. Secondary Outcome: Number of Participants Reporting pIMDs up to the End of Follow-up Study Period (Month 6)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 up to the end of follow-up period (Month 6)
Population: The analysis was performed on the Exposed Set that included all participants who received the study intervention dose.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
Number analyzed (Participants) | 40 | 39 | 43
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 4-day follow-up period after vaccination. Unsolicited AEs were collected during the 30-day follow-up period after vaccination. SAEs and pIMDs were collected throughout the study period (from Day 1 to Month 6).
Arm/Group | High Dose_AS01E Group | Low Dose_AS01E Group | Medium Dose_AS01E Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/39 | 2/43
Other Adverse Events (participants affected / at risk) | 22/40 | 25/39 | 29/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose_AS01E Group (N=40) | Low Dose_AS01E Group (N=39) | Medium Dose_AS01E Group (N=43)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose_AS01E Group (N=40) | Low Dose_AS01E Group (N=39) | Medium Dose_AS01E Group (N=43)
Injection site pain (General disorders) | 21 (21) | 23 (23) | 26 (26)
Injection site erythema (General disorders) | 1 (1) | 6 (6) | 5 (5)
Injection site swelling (General disorders) | 0 (0) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 4 (4)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (3)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sebaceous adenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transferrin saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT04657198/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT04657198/SAP_001.pdf